CLINICAL TRIAL: NCT03200509
Title: Efficacy of a Multimodal Physical Activity Intervention With Supervised Exercises, Health Coaching and an Activity Monitor on Physical Activity Levels of Patients With Chronic Nonspecific Low Back Pain: PAyBACK Trial
Brief Title: Efficacy of a Multimodal Physical Activity Intervention in Patients With Chronic Nonspecific Low Back Pain
Acronym: PAyBACK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Collaborators: University of Sydney (Other)
Responsible Party: Principal Investigator, Crystian Bitencourt Soares de Oliveira, PhD student, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1718
Record Dates: First submitted 2017-06-22; First posted 2017-06-27 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Low Back Pain
Keywords: nonspecific low back pain; chronic pain
MeSH Terms: conditions — Low Back Pain; Chronic Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity Intervention (Experimental): The participants from both groups will receive a group exercise program, including a combination of general, stabilisation, strengthening and resistance exercises. In addition, the intervention group will receive health coaching sessions and an activity monitor.
  Interventions: Other: Physical Activity Intervention
- Control group (Sham Comparator): The participants from both groups will receive a group exercise program, including a combination of general, stabilisation, strengthening and resistance exercises. The participants allocated to the control group will receive sham health coaching and a sham activity monitor, in addition to the exercise program.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Physical Activity Intervention — Participants will receive a group exercise program, health coaching sessions and an activity monitor.
  Arms: Physical Activity Intervention
Other: Control group — Participants will receive a group exercise program, sham health coaching sessions and a sham activity monitor.
  Arms: Control group

SUMMARY:
Physical activity plays an important role in the management of chronic low back pain (LBP). Engaging in an active lifestyle is associated with a better prognosis. Nevertheless, there is evidence to suggest that patients with chronic LBP are less likely to meet recommended physical activity levels. Furthermore, while exercise therapy has been endorsed by recent clinical practice guidelines, evidence from systematic reviews suggests that its effect on pain and disability are at best moderate and not sustained over time. A limitation of current exercises programs for chronic LBP is that these programs are not designed to change patient's behaviour toward an active lifestyle. Therefore, the objective of this study is to investigate the short and long-term efficacy of a multimodal intervention consisting of supervised exercises, health coaching and use of an activity monitor (i.e. Fitbit Flex) compared to supervised exercises plus sham coaching and a sham activity monitor on physical activity levels, pain intensity and disability in patients with chronic nonspecific LBP.

ELIGIBILITY:
Inclusion Criteria:

* Chronic nonspecific LBP, defined as pain and discomfort localised below the costal margin and above the inferior gluteal folds, with or without leg pain and of at least 3 months' duration

Exclusion Criteria:

* Serious spine pathology (e.g. tumors, fractures, and inflammatory diseases)
* Nerve root compromise (i.e. at least 2 of the following signs: weakness, reflex change, or sensation loss associated with the same spinal nerve)
* Spinal surgery
* Pregnancy
* Illiteracy
* Insufficient understanding of the Portuguese language
* Cardiorespiratory Diseases fibromyalgia or any other musculoskeletal condition that may affect activity and movement will be excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-08-15 (Estimated)

PRIMARY OUTCOMES:
Physical activity levels - Counts per minute | Post-intervention (i.e. 3 months after randomisation)
  Counts per minute will be measured with the Actigraph GT3X (ActiGraph, LLC, Pensacola, FL, USA).
Pain intensity | Post-intervention (i.e. 3 months after randomisation)
  Numerical Rating Scale for Pain assessment (NRS) (0-10)
Disability | Post-intervention (i.e. 3 months after randomisation)
  Roland Morris Disability Questionnaire (RMDQ) (0-24)

SECONDARY OUTCOMES:
Physical activity levels - Counts per minute | 6 and 12-month assessment after randomisation
  Counts per minute will be measured with the Actigraph GT3X (ActiGraph, LLC, Pensacola, FL, USA).
Pain intensity | 6 and 12-month assessment after randomisation
  Numerical Rating Scale for Pain assessment (NRS) (0-10)
Disability | 6 and 12-month assessment after randomisation
  Roland Morris Disability Questionnaire (RMDQ) (0-24)
Physical activity levels - light physical activity | Post-intervention (i.e. 3 months after randomisation) and at 6 and 12-month follow-up
  Time spent in light physical activity will be measured with the Actigraph GT3X (ActiGraph, LLC, Pensacola, FL, USA).
Physical activity levels - moderate-to-vigorous physical activity | Post-intervention (i.e. 3 months after randomisation) and at 6 and 12-month follow-up
  Time spent in moderate-to-vigorous physical activity will be measured with the Actigraph GT3X (ActiGraph, LLC, Pensacola, FL, USA).
Physical activity levels - steps | Post-intervention (i.e. 3 months after randomisation) and at 6 and 12-month follow-up
  Number of steps will be measured with the Actigraph GT3X (ActiGraph, LLC, Pensacola, FL, USA).
Sedentary behavior | Post-intervention (i.e. 3 months after randomisation) and at 6 and 12-month follow-up
  Time spent in sedentary behavior will be measured with the Actigraph GT3X (ActiGraph, LLC, Pensacola, FL, USA).
Self-reported physical activity level | Post-intervention (i.e. 3 months after randomisation) and at 6 and 12-month follow-up
  Baecke Habitual Physical Activity Questionnaire
Self-reported sedentary behavior | Post-intervention (i.e. 3 months after randomisation) and at 6 and 12-month follow-up
  Questions about the time spent in sedentary behavior
Depression | Post-intervention (i.e. 3 months after randomisation) and at 6 and 12-month follow-up
  The Center for Epidemiological Studies - Depression (CES-D) scale (0-60)
General quality of life | Post-intervention (i.e. 3 months after randomisation) and at 6 and 12-month follow-up
  EuroQol visual analogue scale (EQ-VAS) (0-100)
Pain self-efficacy | Post-intervention (i.e. 3 months after randomisation) and at 6 and 12-month follow-up
  Pain Self-Efficacy Questionnaire (PSEQ) (0-60)
Weight-related outcomes - Body mass index | Post-intervention (i.e. 3 months after randomisation) and at 6 and 12-month follow-up
  Body mass index
Weight-related outcomes - Waist-to-hip circumference | Post-intervention (i.e. 3 months after randomisation) and at 6 and 12-month follow-up
  Waist-to-hip circumference
Global Perceived Effect Scale (GPES) | Post-intervention (i.e. 3 months after randomisation)
  Perception of recovery

CONTACTS AND LOCATIONS:
Locations (1):
- Sao Paulo State University, Presidente Prudente, São Paulo, Brazil

REFERENCES:
- [Background] Oliveira CB, Franco MR, Maher CG, Tiedemann A, Silva FG, Damato TM, Nicholas MK, Christofaro DGD, Pinto RZ. The efficacy of a multimodal physical activity intervention with supervised exercises, health coaching and an activity monitor on physical activity levels of patients with chronic, nonspecific low back pain (Physical Activity for Back Pain (PAyBACK) trial): study protocol for a randomised controlled trial. Trials. 2018 Jan 15;19(1):40. doi: 10.1186/s13063-017-2436-z. PMID 29334992
- [Derived] Oliveira CB, Christofaro DGD, Maher CG, Franco MR, Tiedemann A, Silva FG, Damato TM, Nicholas MK, Pinto RZ. Adding Physical Activity Coaching and an Activity Monitor Was No More Effective Than Adding an Attention Control Intervention to Group Exercise for Patients With Chronic Nonspecific Low Back Pain (PAyBACK Trial): A Randomized Trial. J Orthop Sports Phys Ther. 2022 May;52(5):287-299. doi: 10.2519/jospt.2022.10874. PMID 35536245
- See also: Physical Activity Interventions for Increasing Objectively Measured Physical Activity Levels in Patients With Chronic Musculoskeletal Pain: A Systematic Review — https://www.ncbi.nlm.nih.gov/pubmed/27111744
- See also: Unlocking the potential of physical activity for back health — https://www.ncbi.nlm.nih.gov/pubmed/28202450